CLINICAL TRIAL: NCT02594384
Title: A Phase 1 Dose Escalation Study of the Safety and Pharmacokinetics of LAM-002A (Apilimod Dimesylate Capsules) Administered Orally in Subjects With Relapsed or Refractory B-Cell Non-Hodgkin's Lymphoma
Brief Title: A Phase I Dose Escalation Study of the Safety and Pharmacokinetics of LAM-002A In Patients With Non-Hodgkin's Lymphoma
Acronym: LAM-002A/NHL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OrphAI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAM-002A-NHL-CLN01
Record Dates: First submitted 2015-10-29; First posted 2015-11-03 (Estimated); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Lymphoma, Non-Hodgkin; Leukemia, Chronic Lymphocytic
Keywords: Phase 1; Safety; Apilimod dimesylate; Pharmacokinetics; Non-Hodgkin Lymphoma; Chronic lymphocytic leukemia
MeSH Terms: conditions — Lymphoma; Leukemia; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — apilimod; Rituximab; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Continuous monotherapy (Experimental): All patients will take LAM-002A two times daily by mouth every day until cancer progression or intolerability.
  Interventions: Drug: LAM-002A
- Intermittent monotherapy (Experimental): All patients will receive LAM-002A at escalating dose levels two times daily by mouth for 3 days on therapy followed by 4 days off therapy every week until cancer progression or intolerability.
  Interventions: Drug: LAM-002A
- LAM-002A + rituximab (Experimental): All patients will receive LAM-002A 125mg two times daily by mouth every day until cancer progression or intolerability and rituximab 375 mg/m2 by vein every week for 4 weeks and then every 8 weeks for 4 times (total of 8 infusions)
  Interventions: Drug: Rituximab
- LAM-002A + atezolizumab (Experimental): All patients will receive LAM-002A 125mg two times daily by mouth every day until cancer progression or intolerability and atezolizumab 1200 mg by vein every 3 weeks until cancer progression or intolerability
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: LAM-002A — 25 mg capsules or 50 mg capsules
  Other Names: apilimod dimesylate
  Arms: Continuous monotherapy; Intermittent monotherapy
Drug: Rituximab — 375 mg/m2 by vein
  Other Names: rituxan
  Arms: LAM-002A + rituximab
Drug: Atezolizumab — 1200 mg by vein
  Other Names: Tecentriq
  Arms: LAM-002A + atezolizumab

SUMMARY:
This is a Phase 1 dose-exploration study of LAM-002A administered by mouth in patients with relapsed or refractory B-cell NHL. Safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD),and preliminary anti-tumor activity will be evaluated.

DETAILED DESCRIPTION:
LAM-002A is supplied as 25-mg or 50-mg capsules and will be administered two times daily or three times daily by mouth in repeated 28-day cycles. Patients will be advised to take the doses at the same time each day.

A 3 + 3 design will be utilized to define a maximum tolerated dose (MTD). The MTD is defined as the highest dose at which no more than 1 of 6 patients (i.e., < 33%) experiences a dose-limiting toxicity (DLT) in the dose cohort.

Once the dose and schedule are established, additional patients will be treated to better characterize the safety, tolerability,PK, PD, and anti-tumor activity of LAM-002A when administered alone or in combination with rituximab or atezolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and comply with the protocol requirements and has signed the informed consent document.
2. Confirmed diagnosis of B-cell Non-Hodgkin's lymphoma limited to follicular lymphoma (FL), diffuse large B-cell lymphoma (DLBCL), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), primary mediastinal B-cell lymphoma (PMBL), or chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) that has progressed and for which standard curative measures do not exist or are no longer effective. Prior therapy must have included a rituximab-based regimen.
3. Patients with DLBCL: Cancer progression after transplant, or be unwilling, unable or not an appropriate candidate for an autologous stem cell or bone marrow transplant
4. Radiographically measurable lymphadenopathy or extranodal lymphoid malignancy (defined as the presence of 1 or more lesions that measure at least 2.0 cm in the longest dimension (as assessed radiographically)
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 2 or less.
6. Adequate organ and marrow function.
7. Able to swallow oral capsules without difficulty.
8. Acceptable birth control.
9. Women of childbearing potential : negative pregnancy test
10. Adequate archival or fresh tumor tissue (from biopsy, bone marrow, or peripheral blood) for analysis of potential predictive biomarkers.

Exclusion Criteria:

1. Patients with central nervous system (CNS) lymphoma are not eligible for the trial unless the disease had been treated and the subject remains without symptoms with no active CNS lymphoma.
2. Not recovered from toxicity due to all prior therapies.
3. Other uncontrolled significant illness.
4. History of malabsorption or other gastrointestinal (GI) disease that may significantly alter the absorption of LAM-002A
5. Major surgery within 28 days prior to first dose of study drug.
6. Past history of tuberculosis (TB) or active infection with TB, human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
7. Lactation or breast feeding.
8. Unable or unwilling to abide by the study protocol or cooperate fully with the Investigator or designee.

This is a shortened list and additional criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-10; Primary Completion 2020-03-09 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Langdon Miller, MD, Study Director — AI Therapeutics
Locations (11):
- United States (11):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Mayo Clinic, Jacksonville, Florida
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - New York University School of Medicine, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Mason Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 12 study centers in the United States, 11 of which enrolled subjects to the trial.
Groups:
- LAM-002A Continuous Monotherapy - 50 mg BID: All participants took 50 mg LAM-002A two times daily by mouth every day until cancer progression or intolerability.
  LAM-002A: 25 mg capsules or 50 mg capsules
- LAM-002A Continuous Monotherapy - 100 mg BID: All participants took 100 mg LAM-002A two times daily by mouth every day until cancer progression or intolerability.
  LAM-002A: 25 mg capsules or 50 mg capsules
- LAM-002A Continuous Monotherapy - 150 mg BID: All participants took 150 mg LAM-002A two times daily by mouth every day until cancer progression or intolerability.
  LAM-002A: 25 mg capsules or 50 mg capsules
- LAM-002A Continuous Monotherapy - 75 mg TID: All participants took 75 mg LAM-002A three times daily by mouth every day until cancer progression or intolerability.
  LAM-002A: 25 mg capsules or 50 mg capsules
- LAM-002A Intermittent Monotherapy - 150 mg BID: All participants received LAM-002A at 150 mg two times daily by mouth for 3 days on therapy followed by 4 days off therapy every week until cancer progression or intolerability.
  LAM-002A: 25 mg capsules or 50 mg capsules
- LAM-002A Continuous Monotherapy - 125 mg: All participants took 125 mg LAM-002A two times daily by mouth every day until cancer progression or intolerability.
  LAM-002A: 25 mg capsules or 50 mg capsules
- LAM-002A + Rituximab: All participants received LAM-002A 125mg two times daily by mouth every day until cancer progression or intolerability and rituximab by vein (IV) every week for 4 weeks and then every 8 weeks for 4 times (total of 8 infusions) or one dose of rituximab IV followed by rituximab subcutaneous (SC) for 3 weeks and then SC every 8 weeks for 4 times (total of 8 doses).
  Rituximab: 375 mg/m^2 IV or rituximab (hyaluronidase) (1,400 mg rituximab and 23,400 Units hyaluronidase human) SC
- LAM-002A + Atezolizumab: All participants received LAM-002A 125mg two times daily by mouth every day until cancer progression or intolerability and atezolizumab 1200 mg by vein every 3 weeks until cancer progression or intolerability
  Atezolizumab: 1200 mg by vein
Period: Overall Study
Arm/Group | LAM-002A Continuous Monotherapy - 50 mg BID | LAM-002A Continuous Monotherapy - 100 mg BID | LAM-002A Continuous Monotherapy - 150 mg BID | LAM-002A Continuous Monotherapy - 75 mg TID | LAM-002A Intermittent Monotherapy - 150 mg BID | LAM-002A Continuous Monotherapy - 125 mg | LAM-002A + Rituximab | LAM-002A + Atezolizumab
Started | 3 | 8 | 5 | 4 | 3 | 20 | 12 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Not Completed | 3 | 8 | 5 | 4 | 3 | 19 | 9 | 7
Not completed — Disease Progression | 3 | 7 | 0 | 2 | 2 | 12 | 5 | 5
Not completed — Adverse Event | 0 | 1 | 4 | 1 | 0 | 6 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Progressive Leukocytosis | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Substantial noncompliance | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set=All subjects who received ≥1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | LAM-002A Continuous Monotherapy - 50 mg BID | LAM-002A Continuous Monotherapy - 100 mg BID | LAM-002A Continuous Monotherapy - 150 mg BID | LAM-002A Continuous Monotherapy - 75 mg TID | LAM-002A Intermittent Monotherapy - 150 mg BID | LAM-002A Continuous Monotherapy - 125 mg | LAM-002A + Rituximab | LAM-002A + Atezolizumab | Total
Number analyzed (Participants) | 3 | 8 | 5 | 4 | 3 | 20 | 12 | 7 | 62
Age, Customized [Count of Participants; unit: Participants]
  Age Category: <65 years | 2 | 3 | 1 | 0 | 0 | 9 | 7 | 2 | 24
  Age Category: ≥65 years | 1 | 5 | 4 | 4 | 3 | 11 | 5 | 5 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 4 | 2 | 2 | 9 | 4 | 3 | 30
  Male | 2 | 3 | 1 | 2 | 1 | 11 | 8 | 4 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 3 | 6 | 4 | 3 | 3 | 16 | 11 | 7 | 53
  Race: Black/African American | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 4
  Race: Other | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic/Latino | 3 | 8 | 5 | 3 | 3 | 16 | 12 | 7 | 57
  Ethnicity: Hispanic/Latino | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 5
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants]
  0, fully active, able to carry on all predisease performance without restrictions | 0 | 5 | 1 | 1 | 1 | 7 | 3 | 0 | 18
  1, restricted in physically strenuous activity but ambulatory and able to do light or sedentary work | 3 | 3 | 3 | 2 | 2 | 11 | 9 | 6 | 39
  2, ambulatory and capable of all self-care but unable to work. Up more than 50% of waking hours | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 4
  3, capable of only limited self-care, confined to bed or chair more than 50% of waking hours | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Maximum Tolerated Dose (MTD) of Continuous Oral LAM-002A
Description: MTD was determined by testing increasing doses up to 125 mg twice a day or 75 mg three times a day orally on dose escalation cohorts with 3 to 6 participants each. In the dose escalation, the cohort sizes of 3 to 6 subjects allow evaluation of regimen safety using a standard definition of MTD (ie, the highest starting dose associated with DLT in <33% of subjects during the first cycle of therapy) when administered continuously (daily administration) and then when administered intermittently (repeated courses of 3 days on and 4 days off).
Time Frame: 28 days
Population: Full analysis set=All subjects who receive ≥1 dose of study drug.
Measure: Number; unit: mg BID
Groups:
- All Participants: All participants who received at least 1 dose of LAM-002A, either at 50 mg BID, 100 mg BID, 150 mg BID, 75 mg TID, or 125 mg BID.
Arm/Group | All Participants
Number analyzed (Participants) | 40
mg BID | 125

2. Secondary Outcome: Peak Plasma Concentration (Cmax) of LAM-002A
Description: Evaluation of the peak plasma concentration (Cmax) of LAM-002A and its metabolites in plasma on Day 1 and Day 8.
Time Frame: 8 days
Population: The PK population included all evaluable subjects who were dosed and had sufficient concentration-time data to estimate ≥1 of the planned PK parameters, as determined by the study pharmacokineticist.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- LAM-002A Continuous Monotherapy - 125 mg BID: All participants took 125 mg LAM-002A two times daily by mouth every day until cancer progression or intolerability.
  LAM-002A: 25 mg capsules or 50 mg capsules
- LAM-002A Intermittent Monotherapy - 150 mg: All participants received LAM-002A at 150 mg two times daily by mouth for 3 days on therapy followed by 4 days off therapy every week until cancer progression or intolerability.
  LAM-002A: 25 mg capsules or 50 mg capsules
Arm/Group | LAM-002A Continuous Monotherapy - 50 mg BID | LAM-002A Continuous Monotherapy - 75 mg TID | LAM-002A Continuous Monotherapy - 100 mg BID | LAM-002A Continuous Monotherapy - 125 mg BID | LAM-002A Continuous Monotherapy - 150 mg BID | LAM-002A Intermittent Monotherapy - 150 mg
Number analyzed (Participants) | 3 | 3 | 8 | 6 | 5 | 3
ng/mL
  Apilimod - Day 1 | 117 (69.6) | 158 (61.6) | 263 (168) | 207 (82.4) | 243 (76.1) | 280 (135)
  Apilimod - Day 8: number analyzed (Participants) | 3 | 3 | 7 | 6 | 2 | 1
  Apilimod - Day 8 | 140 (95.1) | 339 (215) | 331 (273) | 331 (287) | 369 (90.5) | 108
  STA-5908 - Day 1 | 112 (85.0) | 114 (71.6) | 215 (88.6) | 144 (92.5) | 196 (142) | 207 (135)
  STA-5908 - Day 8: number analyzed (Participants) | 3 | 3 | 7 | 5 | 2 | 1
  STA-5908 - Day 8 | 103 (43.7) | 239 (195) | 278 (137) | 234 (173) | 240 (99.7) | 113
  STA-5944 - Day 1 | 209 (145) | 243 (124) | 346 (131) | 281 (125) | 369 (306) | 466 (247)
  STA-5944 - Day 8: number analyzed (Participants) | 3 | 3 | 7 | 5 | 2 | 1
  STA-5944 - Day 8 | 188 (101) | 436 (334) | 439 (215) | 383 (225) | 391 (9.90) | 260
  STA-6048 - Day 1 | 63.2 (40.2) | 59.9 (54.0) | 136 (64.2) | 90.0 (58.6) | 131 (134) | 145 (66.0)
  STA-6048 - Day 8: number analyzed (Participants) | 3 | 3 | 7 | 5 | 2 | 1
  STA-6048 - Day 8 | 60.6 (32.0) | 154 (113) | 161 (43.0) | 122 (81.7) | 116 (87.4) | 140

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of LAM-002A
Description: Evaluation of the Area under the concentration-time curve from time-zero to the time of the last quantifiable concentration (AUClast) of LAM-002ALAM-002A and its metabolites in plasma on Day 1 and Day 8.
Time Frame: 8 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | LAM-002A Continuous Monotherapy - 50 mg BID | LAM-002A Continuous Monotherapy - 75 mg TID | LAM-002A Continuous Monotherapy - 100 mg BID | LAM-002A Continuous Monotherapy - 125 mg BID | LAM-002A Continuous Monotherapy - 150 mg BID | LAM-002A Intermittent Monotherapy - 150 mg BID
Number analyzed (Participants) | 3 | 3 | 8 | 6 | 5 | 3
h*ng/mL
  Apilimod - Day 1 | 238 (88.1) | 583 (290) | 515 (221) | 562 (234) | 700 (290) | 777 (437)
  Apilimod - Day 8: number analyzed (Participants) | 3 | 3 | 7 | 5 | 2 | 1
  Apilimod - Day 8 | 374 (119) | 1040 (483) | 1130 (930) | 1290 (1040) | 1060 (85.7) | 563
  STA-5944 - Day 1 | 542 (214) | 1020 (659) | 1120 (550) | 1180 (587) | 1590 (1420) | 1700 (843)
  STA-5944 - Day 8: number analyzed (Participants) | 3 | 3 | 7 | 5 | 2 | 1
  STA-5944 - Day 8 | 653 (365) | 2070 (1430) | 1810 (1240) | 1860 (1160) | 1320 (211) | 1350
  STA-5908 - Day 1 | 312 (156) | 526 (291) | 762 (371) | 625 (419) | 936 (734) | 968 (547)
  STA-5908 - Day 8: number analyzed (Participants) | 3 | 3 | 7 | 5 | 2 | 1
  STA-5908 - Day 8 | 433 (195) | 1140 (818) | 1360 (796) | 1270 (875) | 1040 (572) | 690
  STA-6048 - Day 1 | 238 (91.2) | 280 (216) | 622 (372) | 443 (325) | 785 (923) | 869 (415)
  STA-6048 - Day 8: number analyzed (Participants) | 3 | 3 | 7 | 5 | 2 | 1
  STA-6048 - Day 8 | 308 (164) | 1040 (780) | 959 (343) | 746 (509) | 556 (397) | 760

4. Secondary Outcome: Objective Response Rate
Description: Anti-tumor response as assessed by investigator according to modified Hallek or Lugano Response Criteria by Disease Type and Cohort
Time Frame: 1 cycle (28 days) up to a maximum of 24 cycles
Population: Full Analysis Set: All participants who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- LAM-002A Intermittent Monotherapy - 150 mg BID: All participants received LAM-002A at escalating dose levels two times daily by mouth for 3 days on therapy followed by 4 days off therapy every week until cancer progression or intolerability.
  LAM-002A: 25 mg capsules or 50 mg capsules
Arm/Group | LAM-002A Continuous Monotherapy - 50 mg BID | LAM-002A Continuous Monotherapy - 100 mg BID | LAM-002A Continuous Monotherapy - 150 mg BID | LAM-002A Continuous Monotherapy - 75 mg TID | LAM-002A Intermittent Monotherapy - 150 mg BID | LAM-002A Continuous Monotherapy - 125 mg | LAM-002A + Rituximab | LAM-002A + Atezolizumab
Number analyzed (Participants) | 3 | 8 | 5 | 4 | 3 | 20 | 12 | 7
Participants
  DLBCL (diffuse large B-cell lymphoma): number analyzed (Participants) | 0 | 4 | 1 | 3 | 1 | 9 | 2 | 4
  DLBCL (diffuse large B-cell lymphoma) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  FL (follicular lymphoma): number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 8 | 8 | 2
  FL (follicular lymphoma) | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 2
  MZL (marginal zone lymphoma): number analyzed (Participants) | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 1
  MZL (marginal zone lymphoma) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  MCL (mantle cell lymphoma): number analyzed (Participants) | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0
  MCL (mantle cell lymphoma) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CLL/SLL (chronic lymphocytic leukemia/ small lymphocytic lymphoma): number analyzed (Participants) | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0
  CLL/SLL (chronic lymphocytic leukemia/ small lymphocytic lymphoma) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0. AEs, including SAEs, were captured from Cycle 1 Day 1 through 30 days after the last dose of study treatment, an average of 4.5 months.
Description: Adverse Events were analyzed for all participants who received at least 1 dose of study treatment.
Arm/Group | LAM-002A Continuous Monotherapy - 50 mg BID | LAM-002A Continuous Monotherapy - 100 mg BID | LAM-002A Continuous Monotherapy - 150 mg BID | LAM-002A Continuous Monotherapy - 75 mg TID | LAM-002A Intermittent Monotherapy - 150 mg BID | LAM-002A Continuous Monotherapy - 125 mg BID | LAM-002A + Rituximab | LAM-002A + Atezolizumab
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/8 | 1/5 | 0/4 | 0/3 | 3/20 | 0/12 | 3/7
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/8 | 1/5 | 2/4 | 0/3 | 9/20 | 5/12 | 6/7
Other Adverse Events (participants affected / at risk) | 3/3 | 8/8 | 5/5 | 4/4 | 3/3 | 20/20 | 12/12 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAM-002A Continuous Monotherapy - 50 mg BID (N=3) | LAM-002A Continuous Monotherapy - 100 mg BID (N=8) | LAM-002A Continuous Monotherapy - 150 mg BID (N=5) | LAM-002A Continuous Monotherapy - 75 mg TID (N=4) | LAM-002A Intermittent Monotherapy - 150 mg BID (N=3) | LAM-002A Continuous Monotherapy - 125 mg BID (N=20) | LAM-002A + Rituximab (N=12) | LAM-002A + Atezolizumab (N=7)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LAM-002A Continuous Monotherapy - 50 mg BID (N=3) | LAM-002A Continuous Monotherapy - 100 mg BID (N=8) | LAM-002A Continuous Monotherapy - 150 mg BID (N=5) | LAM-002A Continuous Monotherapy - 75 mg TID (N=4) | LAM-002A Intermittent Monotherapy - 150 mg BID (N=3) | LAM-002A Continuous Monotherapy - 125 mg BID (N=20) | LAM-002A + Rituximab (N=12) | LAM-002A + Atezolizumab (N=7)
Nausea (Gastrointestinal disorders) | 0 | 3 | 3 | 3 | 0 | 9 | 6 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 2 | 6 | 6 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3 | 3 | 0 | 4 | 3 | 4
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 1 | 3 | 1 | 5
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 4 | 2 | 2 | 1 | 10 | 7 | 1
Asthenia (General disorders) | 0 | 1 | 1 | 0 | 0 | 5 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 0 | 2 | 0 | 3 | 2 | 1
Chills (General disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Eye complication associated with device (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hemoglobin decreased (Investigations) | 0 | 3 | 0 | 2 | 0 | 5 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 2 | 2 | 0 | 0 | 4 | 1 | 0
Platelet count decreased (Investigations) | 0 | 3 | 0 | 1 | 0 | 3 | 2 | 1
Neutrophil count decreased (Investigations) | 0 | 2 | 0 | 1 | 0 | 3 | 2 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Blood phosphorus increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Ammonia increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood lactic acid increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Blood sodium increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 4 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 2 | 1 | 1 | 2 | 3 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asterixis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2
Tooth abscess (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 1 | 4 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 3 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 8 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 2 | 2
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 2 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 4 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 2 | 1 | 2 | 1 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Right ventricular enlargement (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus operation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Participants receiving LAM-002A with a regimen of 125 mg BID were accrued to both dose escalation (N=6) and then dose expansion (N=14), the results for the combined total (N=20) for this group is presented. Additionally, a MTD for the intermittent dosing regimen (3 days on and 4 days off every 7 days) was not established due to the shift of the trial to the dose expansion (monotherapy or combination therapy); the intermittent regimen was not further pursued after 3 subjects had been accrued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT02594384/Prot_SAP_000.pdf